CLINICAL TRIAL: NCT01906788
Title: THE OPTIMAL TIMING OF PRIMAQUINE TO PREVENT MALARIA TRANSMISSION AFTER ARTEMISININ-COMBINATION THERAPY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kilimanjaro Clinical Research Institute (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: PRIMAQUINE STUDY
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Malaria Transmission
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Active Comparator): Active comparator: Artemether Lumefantrine 6 dose regime orally
  Interventions: Drug: Artemether Lumefantrine
- Group 2 (Experimental): Experimental: Artemether Lumefantrine 6 dose regime Plus single dose Primaquine (0.75/kg) on day 0
  Interventions: Drug: Artemether Lumefantrine 6 dose regimen & single dose of Primaquine on day 0
- Group 3 (Experimental): Experimental: Artemether Lumefantrine 6 dose regimen plus single dose of Primaquine (0.75/kg) on day 2
  Interventions: Drug: Artemether Lumefantrine 6 dose regimen and single dose Primaquine on day 2

INTERVENTIONS:
Drug: Artemether Lumefantrine
  Arms: Group 1
Drug: Artemether Lumefantrine 6 dose regimen & single dose of Primaquine on day 0
  Arms: Group 2
Drug: Artemether Lumefantrine 6 dose regimen and single dose Primaquine on day 2
  Arms: Group 3

SUMMARY:
The investigators' Hypothesis is that "The correct timing of gametocytocidal drug in combination with an effective Artemisinin Combination Therapy can limit the infectiousness of malaria-infected individuals to less than one week after initiation of treatment"

DETAILED DESCRIPTION:
Global malaria elimination is back on the agenda, gametocytocidal drugs such as primaquine are currently advocated for use in the interventions that aim to interrupt malaria transmission and hence elimination. Mature gametocytes are responsible for malaria transmission. Artemisinin based combination therapies (ACTs) has limited effect on the young gametocytes. Primaquine is able to clear mature gametocytes that remain after treatment with ACTs. Complete clearance of mature gametocytes will depend on the ideal time primaquine is given after ACT. It is important therefore that is administered at optimal time in order to have significant impact on clearing gametocytes to interrupt malaria transmission. An additional consideration is operational administration of Primaquine and compliance both of which are likely to be enhanced if the drug is administered on the day of diagnosis.

In this study, the investigators aim to determine optimal timing of primaquine administration in addition to ACT by comparing administration on day 0 with administration on day 2.

The investigators' primary end points are gametocyte prevalence and density by microscopy and Quantitative Nucleic Acid Based Amplification (QT-NASBA) on day 14, which will be compared between the two primaquine treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 years - 17 years
* Residents of research area
* Willingness to come for complete scheduled follow-up.
* Uncomplicated malaria with P. falciparum mono-infection
* Axillary temperature > 37.5°C and < 39.5°C, or history of fever in previous 48 hours.
* No history of adverse reactions to study medication
* Understanding of the procedures of the study by parent or guardian and willing to participate by signing written informed consent forms

Exclusion Criteria:

* Haemoglobin below 9g/dl
* Inability to take drugs orally
* Known hypersensitivity to any of the drugs given
* Reported treatment with antimalarial chemotherapy in the past 2 weeks
* Evidence of chronic disease or acute infection other than malaria
* Domicile outside the study area
* Signs of severe malaria( such as respiratory distress, altered consciousness deep breathing, anaemia)
* Participating in other malaria studies conducted in the region
* Mixed malaria parasite species infection
* Positive pregnant test by Urine (UPT) if participant is female aged above 12 years
* G6PD deficient using the fluorescence spot test

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Gametocyte prevalence and density by microscopy and QT-NASBA | Day 14
  By microscopy and QT-NASBA techniques we will determine and compare gametocyte prevalence and density on day 14 between the Primaquine treatment 2 and 3 arms.

SECONDARY OUTCOMES:
Haemoglobin level | days 3, 7, 10 and 14
  We will compare the level of baseline haemoglobin on days 3, 7, 10 and 14 after the start of treatment between the two Primaquine arms

OTHER OUTCOMES:
Proportion of infected mosquitoes | day 7
  We will determine the proportion of infected mosquitoes on day 7 after initiation of treatment and the intensity of infection (oocyst burden)by use of membrane feeding assay technique.

CONTACTS AND LOCATIONS:
Overall Officials: Seif Shekalaghe, MD, PhD, Principal Investigator — Kilimanjaro Clinical Research Institute and Ifakara Health Institute
Locations (1):
- Bagamoyo Research and Training Centre, Bagamoyo, Tanzania

REFERENCES:
- [Derived] Shekalaghe S, Mosha D, Hamad A, Mbaga TA, Mihayo M, Bousema T, Drakeley C, Abdulla S. Optimal timing of primaquine to reduce Plasmodium falciparum gametocyte carriage when co-administered with artemether-lumefantrine. Malar J. 2020 Jan 21;19(1):34. doi: 10.1186/s12936-020-3121-3. PMID 31964380